CLINICAL TRIAL: NCT05982249
Title: Effectiveness of Recorded Hypnosis and Virtual Reality in Patients Undergoing a Bone Marrow Examination at the Hematology Unit
Brief Title: Hypnosis and Virtual Reality in Bone Marrow Examination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0053-23-BNZ
Record Dates: First submitted 2023-07-16; First posted 2023-08-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-07

CONDITIONS: Hematologic Diseases
Keywords: Bone marrow; Procedure; Hematology; Hypnosis; Guided imagery; Virtual reality
MeSH Terms: conditions — Hematologic Diseases | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis (H) (Experimental): Patients will be given earphones to hear a hypnotic script that was recorded by Dr. Zahi Arnon, a psychologist specializing in hypnosis after observing about ten bone marrow (BM) examinations at the hematology institute. The length of the recording is about 7 minutes.
  Interventions: Device: Hypnosis
- Virtual reality (VR) (Experimental): Patients will be connected to a VR device that will transmit to the patient's choice a 3D screen and soothing noise for about 7 minutes.
  Interventions: Device: Virtual reality (VR)
- Control (C) (No Intervention)

INTERVENTIONS:
Device: Hypnosis — Patients will be given earphones to hear a hypnotic script that was recorded by Dr. Zahi Arnon, a psychologist specializing in hypnosis after observing about ten BM examinations at the hematology institute. The length of the recording is about 7 minutes.
  Arms: Hypnosis (H)
Device: Virtual reality (VR) — Patients will be connected to a VR device that will transmit to the patient's choice a 3D screen and soothing noise for about 7 minutes.
  Arms: Virtual reality (VR)

SUMMARY:
The goal of this clinical trial is to compare the effects of hypnosis, virtual reality or their combination in patients undergoing a bone marrow procedure.

The main question it aims to answer is whether such interventions may relieve anxiety and other symptoms described by patients undergoing the procedure.

Before the bone marrow procedure and after being explained on the study and signing informed consent, the nurse will measure vital signs and participants will fill-out a 2-minutes' questionnaire and will be assigned to one of 3 groups:

* Hearing a 7-minutes hypnotic script via earphones
* Seeing and hearing virtual images and sounds via a virtual reality device during 7 minutes
* None of these After these interventions or 10 minutes after assignation for patients not receiving intervention, patients will fill questionnaires again (about 5 minutes for filling the 2 questionnaires) and vital signs will be measured again. Then the bone marrow procedure will be performed. After the bone marrow procedure, the participants will fill-out another 2-minutes questionnaire and vital signs will be measured by the nurse.

Researchers will compare hypnotic script, virtual reality, their combination or none of them to see if they can affect anxiety and other complaints in patients undergoing a bone marrow procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Candidate for a BM examination at the hematology unit
3. Ability to answer questionnaires in Hebrew, Arabic or Russian
4. Informed consent form signing

Exclusion Criteria:

1. Major hearing impairment
2. Major visual impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Symptoms experienced by patients undergoing bone marrow procedure | Through study completion, an average of 1 hour
  Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire: requires participants to nominate one or two concerns and, using a seven-point scale from 0 (worse outcome) to 6 (best outcome), to score these concerns and their general feeling of wellbeing

SECONDARY OUTCOMES:
Absorption, dissociation, immersion and time perception | Through study completion, an average of 1 hour
  Validated questionnaire on absorption, dissociation, immersion and time perception
Sedation | Through study completion, an average of 1 hour
  Type and dose of sedation used during procedure
Use of analgesics | Through study completion, an average of 1 hour
  Type and dose of analgesics
Blood pressure | Through study completion, an average of 1 hour
  Blood pressure
Pulse | Through study completion, an average of 1 hour
  Pulse
Respiratory rate | Through study completion, an average of 1 hour
  Respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Levy Yurkovski, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT05982249/Prot_000.pdf